CLINICAL TRIAL: NCT00806338
Title: A Phase I, Double-Blind, Randomized, Placebo-Controlled Ascending IV Multiple Dose Tolerance and Pharmacokinetic Study of Trodusquemine (MSI-1436) in Obese or Overweight Type 2 Diabetic Volunteers
Brief Title: An Ascending Multi-Dose, Tolerance and Pharmacokinetic Study in Obese or Overweight Type 2 Diabetic Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genaera Corporation (Industry)
Responsible Party: Michael Gast, MD, PhD, Genaera Corporation
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSI-1436C-102
Record Dates: First submitted 2008-01-21; First posted 2008-12-10 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — 3-N-1(spermine)-7, 24-dihydroxy-5-cholestane 24-sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Trodusquemine (MSI-1436) 3mg/m2 (Experimental)
  Interventions: Drug: Trodusquemine (MSI-1436)
- Trodusquemine (MSI-1436) 6mg/m2 (Experimental)
  Interventions: Drug: Trodusquemine (MSI-1436)
- Trodusquemine (MSI-1436) 10mg/m2 (Experimental)
  Interventions: Drug: Trodusquemine (MSI-1436)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trodusquemine (MSI-1436) — A single dose of Trodusquemine (MSI-1436) will be administered every 72 hours on Days 0, 3, 6, 9, 12, 15, 18 and 21. Doses are 3mg/m2 in cohort 1, 6mg/m2 in cohort 2 and 10mg/m2 in cohort 3.
  Arms: Trodusquemine (MSI-1436) 10mg/m2; Trodusquemine (MSI-1436) 3mg/m2; Trodusquemine (MSI-1436) 6mg/m2
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerance of multiple intravenous (through a vein) doses of trodusquemine (MSI-1436) in obese or overweight, type 2 diabetics.

DETAILED DESCRIPTION:
Different amounts of trodusquemine (MSI-1436) will be given to each volunteer group throughout the study. Another purpose is to evaluate the pharmacokinetics (PK - the study of the way the drug enters and leaves the blood and tissues over time) of trodusquemine (MSI-1436). Finally, this study will also determine whether trodusquemine (MSI-1436) has any effect on appetite, mood or behavior, and selective biomarkers (substances in your blood that may change in response to the study drug).

ELIGIBILITY:
Inclusion Criteria:

1. male or female obese or overweight type 2 diabetic subjects, between 18 and 65 years old (inclusive) either treatment naïve or who are inadequately controlled on metformin alone;
2. subjects receiving metformin should be on stable dose for at least two weeks prior to enrollment;
3. have a fasting blood sugar of ≥ 100 mg/dL and hemoglobin A1C ≥ 7.5% (but ≤ 11.0%) at study entry;
4. of any race who are in good health (based on medical history, physical examination, electrocardiograms [ECGs], and clinical laboratory tests);
5. non-smokers (refrained from any tobacco or nicotine usage, including smokeless tobacco, nicotine patches, etc.,) for 6 months prior to Day 0 of the study. Subjects must have cotinine levels below those measured for smokers based on reference lab values;
6. body mass index (BMI) of 27-40 kg/m2;
7. able to execute informed written consent;
8. willingness to remain in the clinic for the inpatient portion of the study and return for follow-up visits as required by the protocol and as deemed necessary by the Principal Investigator;

Exclusion Criteria:

1. likely allergy or sensitivity to any components of Trodusquemine (MSI-1436C) for Injection;
2. any subject with a history of severe allergy or bronchial asthma;
3. a clinically significant history of or current abnormality or disease of any organ system, including renal, hepatic, gastrointestinal, cardiovascular (except hyperlipidemia or controlled hypertension), pulmonary (including chronic asthma), endocrine (except diabetes), central nervous, or hematologic systems, or recent clinically significant surgery;
4. history of seizure, epilepsy, severe head injury, multiple sclerosis, or other known neurological conditions;
5. abnormal pre-admission vital signs, physical examination, clinical laboratory, or any safety variable which is considered clinically significant for this population by the Principal Investigator or Sponsor (or designee). Subjects with an abnormal serum creatinine should not be enrolled. Subjects with AST (SGOT), ALT (SGPT), GGT, alkaline phosphatase, bilirubin, blood urea nitrogen (BUN), prothrombin time (PT), or activated partial thromboplastin time (aPPT) >1.5 times above the upper limit of normal should not be enrolled;
6. any subject with a clinically significant mental or physical illness within 1 year prior to the first dose, including a history of alcohol and/or drug abuse within 1 year prior to the first dose of study medication;
7. Insulin requiring diabetics;
8. any subject who has received any known hepatic or renal clearance altering agents (eg, erythromycin, cimetidine, barbiturates, phenothiazines, St. John's Wort, etc.) within a period of 90 days prior to the first dose of study medication;
9. any subject who has received any approved prescription anti-obesity drug or has taken any over-the-counter medication for weight loss or who has received a thiazolidinedione or exanatide within a period of 90 days prior to the first dose of study medication;
10. ingestion or use of any investigational medication or device within 60 days prior to the first dose of study medication; ingestion or use of any investigational anti-obesity medication is prohibited within 3 months prior to the first dose of study medication;
11. any subject with history of malignancy in last 5 years, with exception of basal and squamous cell carcinomas of the skin;
12. any subject who is positive for HBsAG, Hepatitis C antibody, Hepatitis A IgM, or Human Immunodeficiency Virus (HIV) Viral Serology tests at the screening visit;
13. a positive qualitative urine drug or alcohol test at screening or at check-in;
14. mental capacity is limited to the extent that the subject cannot provide legal consent or understand information regarding the study;
15. any subject who has had a 10% weight loss in the past 3 months prior to the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerance of multiple intravenous doses of trodusquemine (MSI-1436) in obese or overweight type 2 diabetics. Safety will be evaluated by physical exams, vital signs assessments, 12-lead ECGs, clinical lab tests and adverse event profile. | 6 months

SECONDARY OUTCOMES:
Effect on glucose tolerance or glucose/insulin relationships | 6 months
Effect on appetite and food consumption | 6 months
Effect on behavior and mood | 6 months
Effect on exploratory biomarkers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kipnes, MD, Principal Investigator — dgd Research; Gilbert Weiner, D.O. AOBFP, Principal Investigator — Cetero Research, San Antonio
Locations (2):
- United States (2):
  - Cetero Research, Miami Gardens, Florida
  - dgd Research, San Antonio, Texas